CLINICAL TRIAL: NCT02999048
Title: Clinical Study on the Treatment of Hypertensive Cerebral Hemorrhage With Panax Notoginseng Saponins
Brief Title: Clinical Study on the Treatment of Hypertensive Intracerebral Hemorrhage With Panax Notoginseng Saponin
Acronym: CSTHIHPNS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The First People's Hospital of Jingzhou (Other)
Responsible Party: Principal Investigator, Zhijian Luo, deputy chief physician, neurology physician, The First People's Hospital of Jingzhou
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012CC47
Record Dates: First submitted 2016-12-13; First posted 2016-12-21 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Hematoma Absorption and Neurological Function Recovery
Keywords: panax notoginseng saponins; hypertensive intracerebral hemorrhage; hematoma; neurological function
MeSH Terms: conditions — Intracranial Hemorrhage, Hypertensive; Hematoma | interventions — xuesetong

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (No Intervention): Patients in the control group received conventional therapy for 17 days.conventional therapy consists of: (1) dehydration therapy by 20%mannitol (Tianjin Bane Medical Drugs Ltd., Co., China.) with the dosage from 125 to 250 ml every 8 h for 7 days depending on their clinically presumed intracranial pressure, (2) therapy to deal with complications including glucose-lowering treatment for hyperglycemia, antihypertensive treatment for hypertension, anti-inflammatory treatment for infection, acid inhibitor for peptic ulcer, and (3) supportive therapy, such as physical cooling, nutritional support, fluid, and electrolyte balance, which was provided as needed.
- intervention group (Other): Patients in the intervention group received the same conventional therapy as in the control group for 3 days, brain CT was re-scanned at the 4th day, and was then given conventional therapy plus XUESAITONG Injection,which was mainly composed of Panax notoginseng saponins for 14 days from the 4th day.
  Interventions: Drug: Panax Notoginseng Saponins

INTERVENTIONS:
Drug: Panax Notoginseng Saponins — Panax Notoginseng Saponins integrated with conventional therapy
  Other Names: XUESAITONG Injection
  Arms: intervention group

SUMMARY:
The purpose of this study is to determine whether panax notoginseng saponins are effective in the treatment of Hypertensive Intracerebral Hemorrhage Patients.

DETAILED DESCRIPTION:
Patients with HICH were randomly assigned to receive either PNS integrated with conventional therapy. Patients were treated with conventional therapy for 3 days, then plus PNS for 14 days. Patients in the control group received conventional therapy for 17days. Hematoma volume measured by CT scanning, National Institutes of Health Stroke Scale (NIHSS) scores, Barthel index (BI), all the three were used to evaluate the therapeutic effect for both groups after two weeks of intervention.

ELIGIBILITY:
Inclusion Criteria:

* with a history of hypertension treated with medication and blood pressure management ( a systolic blood-pressure target of 140 to 179 mmHg and a diastolic blood-pressure target of 70 to 100 mmHg) during the period of hospitalization,
* the site of hematoma located in one of the cerebral hemispheres,
* hematoma volume 10-30ml,
* no blood in the ventricles,
* within 24 hours of onset of first-time acute intracerebral hemorrhage,
* no loss of consciousness (drowsiness acceptable).

Exclusion Criteria:

* cerebellar or brainstem hemorrhage,
* intracerebral hemorrhage caused by bleeding diathesis, aneurysms, vascular malformations, improperly using anticoagulant drugs, or suspicious amyloid angiopathy,
* subarachnoid hemorrhage; multifocal hemorrhage,
* mixed stroke or hemorrhagic infarct,
* coexisting systematic diseases such as heart or kidney failure, tumors, gastrointestinal hemorrhage and so on,
* pregnant or lactating women,
* a history of XUESAITONG injection anaphylaxis.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Hematoma volume | within the 14 days after two weeks of intervention
National Institutes of Health Stroke Scale (NIHSS) scores | within the 14 days after two weeks of intervention
  were measured for stroke severity
Barthel index | within the 14 days after two weeks of intervention
  were measured for quality of life

SECONDARY OUTCOMES:
adverse events | 14 days
  such as rash, allergic shock

REFERENCES:
- [Result] Cheung RT. Update on medical and surgical management of intracerebral hemorrhage. Rev Recent Clin Trials. 2007 Sep;2(3):174-81. doi: 10.2174/157488707781662751. PMID 18474003
- [Result] Nilsson OG, Lindgren A, Brandt L, Saveland H. Prediction of death in patients with primary intracerebral hemorrhage: a prospective study of a defined population. J Neurosurg. 2002 Sep;97(3):531-6. doi: 10.3171/jns.2002.97.3.0531. PMID 12296635
- [Result] Zhao X, Wang Y, Wang C, Li S, Wang Y, Yang Z. Quantitative evaluation for secondary injury to perihematoma of hypertensive cerebral hemorrhage by functional MR and correlation analysis with ischemic factors. Neurol Res. 2006 Jan;28(1):66-70. doi: 10.1179/016164106X91898. PMID 16464365
- [Result] Kang DW, Han MK, Kim HJ, Yun SC, Jeon SB, Bae HJ, Kwon SU, Kim JS. New ischemic lesions coexisting with acute intracerebral hemorrhage. Neurology. 2012 Aug 28;79(9):848-55. doi: 10.1212/WNL.0b013e3182648a79. Epub 2012 Jul 25. PMID 22843271
- [Result] Li JY, Yuan LX, Zhang GM, Zhou L, Gao Y, Li QB, Chen C. Activating blood circulation to remove stasis treatment of hypertensive intracerebral hemorrhage: A multi-center prospective randomized open-label blinded-endpoint trial. Chin J Integr Med. 2016 May;22(5):328-34. doi: 10.1007/s11655-016-2467-7. Epub 2016 Apr 30. PMID 27338955
- [Result] Chen X, Zhou M, Li Q, Yang J, Zhang Y, Zhang D, Kong S, Zhou D, He L. Sanchi for acute ischaemic stroke. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD006305. doi: 10.1002/14651858.CD006305.pub2. PMID 18843711
- [Result] Zhang X, Wu J, Zhang B. Xuesaitong injection as one adjuvant treatment of acute cerebral infarction: a systematic review and meta-analysis. BMC Complement Altern Med. 2015 Feb 27;15:36. doi: 10.1186/s12906-015-0560-4. PMID 25888429
- [Result] Kim CH, Kim JS. Development of cerebral infarction shortly after intracerebral hemorrhage. Eur Neurol. 2007;57(3):145-9. doi: 10.1159/000098465. Epub 2007 Jan 10. PMID 17213720
- [Result] Nyquist P. Management of acute intracranial and intraventricular hemorrhage. Crit Care Med. 2010 Mar;38(3):946-53. doi: 10.1097/CCM.0b013e3181d16a04. PMID 20068459
- [Result] Wasserman JK, Zhu X, Schlichter LC. Evolution of the inflammatory response in the brain following intracerebral hemorrhage and effects of delayed minocycline treatment. Brain Res. 2007 Nov 14;1180:140-54. doi: 10.1016/j.brainres.2007.08.058. Epub 2007 Sep 5. PMID 17919462
- [Result] Sun K, Wang CS, Guo J, Liu YY, Wang F, Liu LY, He JG, Fan JY, Han JY. Effect of Panax notoginseng saponins on lipopolysaccharide-induced adhesion of leukocytes in rat mesenteric venules. Clin Hemorheol Microcirc. 2006;34(1-2):103-8. PMID 16543624
- [Result] Wang YX, Yan A, Ma ZH, Wang Z, Zhang B, Ping JL, Zhu JS, Zhou Y, Dai L. Nuclear factor-kappaB and apoptosis in patients with intracerebral hemorrhage. J Clin Neurosci. 2011 Oct;18(10):1392-5. doi: 10.1016/j.jocn.2010.11.039. Epub 2011 Jul 22. PMID 21782444
- [Result] Li H, Deng CQ, Chen BY, Zhang SP, Liang Y, Luo XG. Total saponins of Panax notoginseng modulate the expression of caspases and attenuate apoptosis in rats following focal cerebral ischemia-reperfusion. J Ethnopharmacol. 2009 Jan 30;121(3):412-8. doi: 10.1016/j.jep.2008.10.042. Epub 2008 Nov 18. PMID 19059471